CLINICAL TRIAL: NCT03123445
Title: The Efficacy and Safety of Continuous Administration of Endostar Combined With Chemotherapy for Patients With Advanced no Small Cell Lung Cancer: An Open-label, no Randomized Controlled Multicenter Phase II Study
Brief Title: Endostar First-line Treatment of Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Shengjing Hospital (Other); General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology,The First Hospital of China Medical University Affiliation: China Medical University, China, China Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOG1701
Record Dates: First submitted 2017-04-05; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: endostar
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — endostar protein; Endostatins; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endostar + Gemcitabine and Cisplatin (Experimental): Patients in this group will be given endostar combined with gemcitabine and cisplatine.
  Interventions: Drug: Endostar; Drug: Gemcitabine; Drug: Cisplatin
- Gemcitabine and Cisplatin (Active Comparator): Patients in this group will be given gemcitabine and cisplatine.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Endostar — Endostar,30mg continuous intravenous injection pump, d1-d7,21 days as one cycle, 4 cycles in total
  Other Names: Recombinant Human Endostatin Injection
  Arms: Endostar + Gemcitabine and Cisplatin
Drug: Gemcitabine — Gemcitabine,1000mg/m2, i.v, d1 and d8 in each cycle, 21 days as one cycle, 4 cycles in total
Drug: Cisplatin — Cisplatin,75mg/m2, i.v, d1 in each cycle, 21 days as one cycle, 4 cycles in total

SUMMARY:
Explore the efficacy and safety of the treatment of Endostar continuous intravenous injection pump combined GP（gemcitabine+cisplatin） scheme for first-line advanced non small cell lung cancer and maintenance treatment.

DETAILED DESCRIPTION:
Explore the efficacy and safety of the treatment of Endostar continuous intravenous injection pump combined GP（gemcitabine+cisplatin） scheme for first-line advanced non small cell lung cancer and maintenance treatment.

main objectives: PFS (progression-free survival) the secondary goal: ORR (overall response rate), DCR (disease control rate) and OS（overall survival）

ELIGIBILITY:
Inclusion Criteria:

* Cytological and histological confirmation（Do not accept single sputum cytology in the diagnosis of patients） in patients diagnosed of lung squamous carcinoma; According to a new IASLC (International Association for the Study of Lung Cance) 2009 lung cancer TNM (tumor node metastasis) stages judged stage IIIB or IV non-small cell lung cancer.
* Must have at least one evaluated lesion,according to the RECIST version 1.1 standard (the longest diameter on spiral CT at least 10 mm,the longest diameter on plain CT at least 20 mm);
* Male or female, age between 18 and 75 years old ;
* ECOG(Eastern Cooperative Oncology Group) PS (performance status ) 0~1；
* Expected survival period ≥ 3 months or more
* Enough blood function: absolute neutrophil count (ANC)≥2 x 109 / L and the platelet count≥ 100 x 109 / L and hemoglobin ≥9 g/dL;
* Enough liver function: total bilirubin acuities≤the upper limit of normal (ULN); aspartate aminotransferase(AST) and Alanine aminotransferase(ALT) acuities ≤2.5 times of the upper limit of normal (ULN); Alkaline phosphatase ≤5 times of the upper limit of normal(ULN);
* Enough renal function：serum creatinine ≤the limit of normal(ULN) or calculated creatinine clearance≥60 mL/min.
* The electrocardiogram (ecg) basically normal,the body had no to heal wounds
* No previous anti-tumor drug therapy, or only received for non metastatic tumor of adjuvant or neoadjuvant chemotherapy, but has ended more than six months before the study start.
* Patients had surgery before,but have more than 4 weeks before the study start, and the patient has recovered;
* Women with completed uterus before intact in the group within 28 days must have a negative pregnancy test results (unless amenorrhea for 24 months). If the pregnancy test from the first time for more than 7 days,the patients need for urine pregnancy test(within 7 days before the first delivery).
* Prior to biological agents, especially e. coli genetically engineered products without severe allergic reactions;
* Sign the informed consent.

Exclusion Criteria:

* Pregnancy, nursing mothers, or female patients with fertility but no contraception.
* Existing serious acute infection, and can not be controlled; Or with fester sex and chronic infection,or wound in delay;
* Original serious heart disease, including: congestive heart failure, uncontrolled high risk arrhythmia, unstable angina, myocardial infarction, severe valvular heart disease, and resistant hypertension;
* With uncontrolled nerve, mental illness or mental disorders, compliance is poor, can't cooperate and response to treatment; Uncontrolled primary brain tumors or central nervous system(CNS) metastases illness, with obvious symptoms in cranial hypertension or nerve spirit;
* With a bleeding tendency
* Researchers believe that patients should not participate in this test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Time Frame: up to month 36
  PFS is a tumor progression or death time of a patient who has an objective record on the date of enrollment. PFS calculation end if the patient was lost, unknown death , or other anti tumor therapy was used.

SECONDARY OUTCOMES:
ORR | Time Frame: change from Baseline at the week 6, 12 of the treatment phase, the month 3, 6, 9 and 12, 15, 18, 21, 24, 27, 30 ,33,36 of the followup phase.
  overall remission rate

CONTACTS AND LOCATIONS:
Overall Officials: liu yunpeng, PhD, Principal Investigator — First Hospital of China Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang J, Gu LJ, Fu CX, Cao Z, Chen QY. Endostar combined with chemotherapy compared with chemotherapy alone in the treatment of nonsmall lung carcinoma: A meta-analysis based on Chinese patients. Indian J Cancer. 2014 Mar;51 Suppl 3:e106-9. doi: 10.4103/0019-509X.154099. PMID 25818734
- [Background] Hu W, Fang J, Nie J, Dai L, Zhang J, Chen X, Ma X, Tian G, Wu D, Han S, Han J, Wang Y, Long J. Efficacy and safety of extended use of platinum-based doublet chemotherapy plus endostatin in patients with advanced nonsmall cell lung cancer. Medicine (Baltimore). 2016 Jul;95(28):e4183. doi: 10.1097/MD.0000000000004183. PMID 27428214
- [Background] Rong B, Yang S, Li W, Zhang W, Ming Z. Systematic review and meta-analysis of Endostar (rh-endostatin) combined with chemotherapy versus chemotherapy alone for treating advanced non-small cell lung cancer. World J Surg Oncol. 2012 Aug 24;10:170. doi: 10.1186/1477-7819-10-170. PMID 22917490
- [Result] Zhang FL, Gao EY, Shu RB, Wang H, Zhang Y, Sun P, Li M, Tang W, Jiang BQ, Chen SQ, Cui FB. Human Recombinant Endostatin Combined with Cisplatin Based Doublets in Treating Patients with Advanced NSCLC and Evaluation by CT Perfusion Imaging. Asian Pac J Cancer Prev. 2015;16(15):6765-8. doi: 10.7314/apjcp.2015.16.15.6765. PMID 26434908